CLINICAL TRIAL: NCT01334736
Title: A Study of Novel Smoking Cessation Interventions in Current and Former Injection Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: TD-10-002
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Dependence
Keywords: smoking cessation; contingency management; spirometry; lung age
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual care (Placebo Comparator)
  Interventions: Behavioral: Usual care
- Lung Age (Active Comparator)
  Interventions: Behavioral: Lung age
- Contingency Management (Active Comparator)
  Interventions: Behavioral: Contingency Management
- Lung age + Contingency Management (Active Comparator)
  Interventions: Behavioral: Lung age + Contingency Management

INTERVENTIONS:
Behavioral: Usual care — After participants have completed the data collection portion of the SHIELD visit, the research assistant will provide the participant with an informational flyer regarding the risks of tobacco smoking and benefits of tobacco cessation. The participant will be provided the phone number for the Tobacco Quit Line in Maryland as well as a list of local tobacco cessation programs. Any questions will be answered by the research assistant. If the participant inquires about nicotine replacement therapy, they will be advised to contact their primary care provider to discuss potential therapeutic options. Spirometry results will be verbally disclosed to participants describing their lung function as a percent of predicted value. A handout with these results will be given to participants. At each follow-up visit, after obtaining CO and questionnaire data, spirometry results will be reviewed and participants will be offered the informational flyer and quit line number.
  Arms: Usual care
Behavioral: Lung age — For individuals randomized to spirometric lung age intervention, after completion of data collection, CO level and acceptable spirometry, the participant will be verbally informed of spirometric results. It will be explained that lung function normally reduces with age and that smoking can damage lung as if they were aging more rapidly than normal using visual depictions. Their lung function estimates based on their chronological age and lung age will be provided. They will be informed that smoking cessation would slow the aging of their lungs. After questions are answered, the participant will receive a written report that includes enumeration of their lung age and chronological age. At initial and follow-up visits, the research assistant will provide the participant with the same informational flyer and Tobacco Quit Line in Maryland as the usual care intervention.
  Arms: Lung Age
Behavioral: Contingency Management — For individuals randomized to CM, after completion of data collection, it will be explained to the participant that they will receive monetary compensation for biological confirmation of tobacco cessation. At each visit, exhaled carbon monoxide levels will be checked. If the subject has a negative CO level, they will be compensated. If a participant has a CO consistent with recent tobacco use, (s)he will receive the payment for attending the visit, but no additional payment at that visit. Spirometry results will be verbally disclosed to participants describing their lung function as a percent of predicted value. A handout with these results will be given to participants. At each follow-up visit, after obtaining CO and questionnaire data, spirometry results will be reviewed and participants will be offered the informational flyer and quit line number.
  Arms: Contingency Management
Behavioral: Lung age + Contingency Management — For individuals randomized to the combined contingency management + spirometric lung age intervention, after completion of data collection, CO level and acceptable spirometry, the participant will be described the process of contingency management as outlined above. Following this, the research assistant will then describe lung age to the participant as described above. At the end of this process, the participant will then receive the informational flyer, quit line and local tobacco cessation program information similar to the usual care intervention. At each follow-up visit, after obtaining CO level and questionnaire outcomes, appropriate CM payment, review of participant's baseline lung age and informational flyer will occur.
  Arms: Lung age + Contingency Management

SUMMARY:
Cigarette smoking is very common in current and former injection drug users and is known to cause chronic lung diseases. Quitting smoking is proven to improve the health of people addicted to cigarettes. . Little information exists regarding the perceptions and characteristics of drug users regarding quitting smoking. Additionally, most programs designed to help people quit smoking are not very successful. One reason these programs may not work well is because it is difficult to motivate people to quit smoking. New methods of motivating changes in behavior include small monetary payments for healthy behavior and reporting breathing tests with the concept of "lung age," which is the age of an average healthy person with similar breathing test results. For example, a health care provider can report results as "Although you are 50 years old, you have the lungs for a 70 year old". In this proposal, the investigators plan to first explore the beliefs and characteristics of current and former injection drug users and how they are related to quitting smoking. The investigators then plan to study whether the use of two new methods of motivation increases the chances that this group will stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker

Exclusion Criteria:

* Enrollment in smoking cessation protocol
* Current use of nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Biologically confirmed tobacco cessation | 6 months
  The primary outcome will be validated tobacco cessation at 6 months. Biologically confirmed tobacco cessation will be assessed by self-report of smoking status combined with CO measurement.

SECONDARY OUTCOMES:
Self efficacy and intention to quit | 6 months
  Self-efficacy and intention to quit smoking will be assessed at baseline using a modified version of the Prochaska stages of change questionnaire. Quit attempts will be enumerated at follow-up visits by asking participants how many quit attempts they made in the prior six months.
Cessation attempts | 6 months
  Cessation attempts will be quantified as the number of sustained cessation attempts lasting more than 7 days, number of sustained cessation attempts lasting more than one month and number of daily cigarettes smoked.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins ALIVE Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Drummond MB, Astemborski J, Lambert AA, Goldberg S, Stitzer ML, Merlo CA, Rand CS, Wise RA, Kirk GD. A randomized study of contingency management and spirometric lung age for motivating smoking cessation among injection drug users. BMC Public Health. 2014 Jul 28;14:761. doi: 10.1186/1471-2458-14-761. PMID 25074396